CLINICAL TRIAL: NCT01332396
Title: Drug Use Investigation for TYKERB Tablet (All Case Investigation)
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: 113092
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients prescribed TYKERB: Patients with HER2 overexpressing inoperable or recurrent breast cancer
  Interventions: Drug: Lapatinib

INTERVENTIONS:
Drug: Lapatinib

SUMMARY:
Data on the safety and efficacy of TYKERB shall be collected from the patients in order to grasp the actual conditions of post-marketing use and assess background information on the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HER2 overexpressing inoperable or recurrent breast cancer

Exclusion Criteria:

* Patients with hypersensitivity to lapatinib or any components
* Pregnant women and women suspected of being pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have "HER2 overexpressing inoperable or recurrent breast cancer" and have received TYKERB for the first time
Sampling Method: Probability Sample
Enrollment: 4054 (Actual)
Dates: Start 2009-06; Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events in Japanese patients treated with TYKERB based on prescribing information under the conditions of general clinical practice | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals